CLINICAL TRIAL: NCT00935948
Title: Phase 3 Clinical Trial - Efficacy and Safety Evaluation of the Drug Imescard Compound Water Smartweed, Adrenalin and Hamamelis Ointment
Brief Title: Efficacy and Safety Evaluation of the Imescard Compound Water Smartweed Ointment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Paulo Dornelles Picon, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04497
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Hemorrhoidal Disease
Keywords: hemorrhoids; hemorrhoidal disease; water smartweed; hamamelis; RCT
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imescard ointment (Active Comparator)
  Interventions: Drug: Imescard compound water smartweed ointment
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imescard compound water smartweed ointment — Patients in this arm were instructed to apply the ointment after waking up, after evacuations and before bedtime, for 5 days.
  Other Names: Imescard; Water smartweed ointment
  Arms: Imescard ointment
Drug: Placebo — Patients in this arm received placebo, with the exact same appearance of the Imescard ointment, and were instructed to apply it at the same intervals and period.
  Arms: Placebo

SUMMARY:
The aim of our study was to assess the clinical efficacy and safety of the drug Imescard compound water smartweed, adrenalin and hamamelis ointment in the treatment of hemorrhoidal disease in adults, in a randomized, double-blind, placebo-controlled clinical trial.

DETAILED DESCRIPTION:
The drug Imescard compound water smartweed ointment is currently registered at the brazilian National Sanitary Surveillance Agency (ANVISA) as a topic hemorrhoidal treatment. It's composed by adrenalin, which produces vasoconstriction, benzocaine, an anesthetic, hamamelis, which is believed to have a desiccative and astringent activity, and water smartweed (Polygonum hydropiperoides), commonly used in the treatment of this condition, with, however, little or no evidence other than tradition to support its use. The aim of this study was to assess the clinical efficacy and safety of this drug in the treatment of hemorrhoidal disease in adults, in a randomized, double-blind, placebo-controlled clinical trial.

Sixty healthy volunteers with ages between 18 to 70 years old who presented with 2nd to 4th degree hemorrhoids were enrolled after clinical and laboratory evaluation (day 0) and then randomized (day 1) to receive either the Imescard ointment after waking up, after evacuations and before bedtime, for 5 days, or placebo, with the exact same appearance and posology. At followup (day 8), patients underwent new clinical and laboratory evaluation. Main outcome was the percentage of patients with 50% improval of symptoms, assessed by a diary containing symptom questionnaires concerning every day of treatment. Secondary outcomes were mean scores of the symptom questionnaires, life quality improval assessed by WHOQOLbrief at days 1 and 8 and adverse effects evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* 2nd to 4th degree hemorrhoids clinically diagnosed
* Proper anticonception, in the case of women in fertile age
* Possibility to abstain from any other drugs (except in emergencies, in wich case the responsible party must be informed)
* Good understanding and agreement to informed consent form

Exclusion Criteria:

* Hypersensitivity to any of the components of the drug
* Use of alcohol or drugs
* Clinical evidence of immunosupression
* Abnormalities in baseline laboratory exams
* Diagnosis of any acute disease in current activity or chronic disease uncontrolled

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Improval of 50% or more in hemorrhoidal symptoms, assessed by questionnaires concerning pain, swelling, secretion and bleeding of hemorrhoids, contained in a diary that patients were instructed to fulfill daily during the treatment. | Days 1 to 5.

SECONDARY OUTCOMES:
Mean scores of the symptom questionnaires mentioned above. | Days 1 to 5.
Life quality was assessed through the questionnaire WHOQOLbrief, at baseline and followup. | Days 1 and 8.
Adverse effects were assessed through a specific field in the diary and at followup during clinical evaluation. | Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil